CLINICAL TRIAL: NCT04391387
Title: Clinical Impact of Different Duration Prone Postition Treatment for Patients With ARDS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chien-Wei Hsu, attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS109-084
Record Dates: First submitted 2020-04-10; First posted 2020-05-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Oxygenation; Driving Pressure
Keywords: acute respiratory distress syndrome; mechanical ventilation; oxygenation; prone position; protective lung ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16-hour prone position (Active Comparator): measure vital signs, PaO2/FiO2, driving pressure one hour before prone position and 1-hour, 8-hour, 16-hour after prone position
  Interventions: Procedure: prone position
- 24-hour prone position (Experimental): measure vital signs, PaO2/FiO2, driving pressure one hour before prone position and 1-hour, 8-hour, 16-hour, 24- hour after prone position
  Interventions: Procedure: prone position

INTERVENTIONS:
Procedure: prone position — a position with the patient lying face down with arms bent comfortably at the elbow and padded with the armboards positioned forward

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a life-threatening disease, patients with ARDS usually need mechanical ventilation. The treatment of ARDS include low tidal volume ventilation, steroid, extracorporeal membraneous oxygenator, inhaled nitric oxide or prone position . Some studies showed prone position had beneficial effect of oxygenation and mortality for severe ARDS patients, the duration of prone position should be at least 10 hours. It is unknown the optimal duration of prone position which is better for severe ARDS patients. This study will compare the clinical differences of 16-hour and 24-hour prone position for severe ARDS patients.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study. All severe ARDS patients were eligible for screening from January 2020 to December 2022. Inclusion criteria include: Patient above 20 year-old with diagnosis of severe ARDS under protective lung ventilation( tidal volume 4-8 ml/kg, plateau pressure < 30cm H2O、PaO2/FiO2 < 150 mmHg、PEEP ≥ 5 cmH2O、FiO2 > 60%）. Patients were excluded if patients were not intubated and mechanically ventilated or contraindication for prone position ventilation (intracranial hemorrhage, massive hemoptysis, unstable hemodynamic status, recent pacemaker implantation, severe facial laceration, open abdominal wound, spine, femur or pelvis fracture or pregnancy). Patients will divide into 2 groups, one is patients supported by 16-hour prone position; another group is patients with 24-hour prone position, each group enrolled 30 patients. The medical records of these patients were analyzed for age, gender, body weight, diagnosis, pulmonary or extrapulmonary ARDS, acute physiology and chronic health evaluation (APACHE) Ⅱscore, days between ARDS to prone position, ICU day, hospital day, ventilator day, pre and post prone position vital signs, laboratory data including arterial blood gas, lactate, respiratory parameters included PaO2/FiO2, peak inspiratory pressure, positive end-expiratory pressure, ventilator mode, steroid treatment, complications (tube dislodge, pressure sore, infection), and mortality outcomes.

The primary endpoint is the difference of oxygenation (PaO2/FiO2), the secondary endpoint are other respiratory parameters, vital signs, ICU day, hospital day, ventilator day, complications and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 20 year-old with diagnosis of severe ARDS under protective lung ventilation (tidal volume 4-8 ml/kg, plateau pressure < 30cm H2O、PaO2/FiO2 < 150 mmHg、PEEP ≥ 5 cmH2O、FiO2 > 60%).

Exclusion Criteria:

* Patients were not intubated and mechanically ventilated or contraindication for prone position ventilation (intracranial hemorrhage, massive hemoptysis, unstable hemodynamic status, recent pacemaker implantation, severe facial laceration, open abdominal wound, spine, femur or pelvis fracture or pregnancy).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
oxygenation | Change from baseline PaO2/FiO2 at 24-hour after prone position
  PaO2/FiO2

SECONDARY OUTCOMES:
respiratory parameters | Change from baseline driving pressure at 24-hour after prone position
  driving pressure
vital sign | Change from baseline driving pressure at 24-hour after prone position
  blood pressure
duration of stay | up to 3 months
  length of ICU stay
complication | up to 3 months
  sliding out of tube
survival | one year
  survival or death

CONTACTS AND LOCATIONS:
Overall Officials: Chien Wei Hsu, MD, Principal Investigator — Kaohsiung VGH
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Result] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Result] Sweeney RM, McAuley DF. Acute respiratory distress syndrome. Lancet. 2016 Nov 12;388(10058):2416-2430. doi: 10.1016/S0140-6736(16)00578-X. Epub 2016 Apr 28. PMID 27133972
- [Result] Alessandri F, Pugliese F, Ranieri VM. The Role of Rescue Therapies in the Treatment of Severe ARDS. Respir Care. 2018 Jan;63(1):92-101. doi: 10.4187/respcare.05752. Epub 2017 Oct 24. PMID 29066591
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Drahnak DM, Custer N. Prone Positioning of Patients With Acute Respiratory Distress Syndrome. Crit Care Nurse. 2015 Dec;35(6):29-37. doi: 10.4037/ccn2015753. PMID 26628543
- [Result] Lee JM, Bae W, Lee YJ, Cho YJ. The efficacy and safety of prone positional ventilation in acute respiratory distress syndrome: updated study-level meta-analysis of 11 randomized controlled trials. Crit Care Med. 2014 May;42(5):1252-62. doi: 10.1097/CCM.0000000000000122. PMID 24368348
- [Result] Fan E, Del Sorbo L, Goligher EC, Hodgson CL, Munshi L, Walkey AJ, Adhikari NKJ, Amato MBP, Branson R, Brower RG, Ferguson ND, Gajic O, Gattinoni L, Hess D, Mancebo J, Meade MO, McAuley DF, Pesenti A, Ranieri VM, Rubenfeld GD, Rubin E, Seckel M, Slutsky AS, Talmor D, Thompson BT, Wunsch H, Uleryk E, Brozek J, Brochard LJ; American Thoracic Society, European Society of Intensive Care Medicine, and Society of Critical Care Medicine. An Official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine Clinical Practice Guideline: Mechanical Ventilation in Adult Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 May 1;195(9):1253-1263. doi: 10.1164/rccm.201703-0548ST. PMID 28459336
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Beitler JR, Shaefi S, Montesi SB, Devlin A, Loring SH, Talmor D, Malhotra A. Prone positioning reduces mortality from acute respiratory distress syndrome in the low tidal volume era: a meta-analysis. Intensive Care Med. 2014 Mar;40(3):332-41. doi: 10.1007/s00134-013-3194-3. Epub 2014 Jan 17. PMID 24435203
- [Result] Tonelli AR, Zein J, Adams J, Ioannidis JP. Effects of interventions on survival in acute respiratory distress syndrome: an umbrella review of 159 published randomized trials and 29 meta-analyses. Intensive Care Med. 2014 Jun;40(6):769-87. doi: 10.1007/s00134-014-3272-1. Epub 2014 Mar 26. PMID 24667919
- See also: Valera, S. (2017). Mobilizing the ECMO patients: Prone positioning during venovenous extracorporeal membrane Oxygenation (vv ECMO). In C. Mossadegh & A. Combes (Eds.), Nursing care and ECMO (pp. 75-82). Cham, Switzerland: Springer. — https://link.springer.com/chapter/10.1007/978-3-319-20101-6_7